CLINICAL TRIAL: NCT02168348
Title: Impact of Malnutrition on the Healing of Foot Lesions in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUILLET 2013
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients With Type 1 or 2 Diabetes; Lesion Situated on a Toe or on the Plantar or Dorsal Side of the Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Diabetic patients with a lesion on the foot
  Interventions: Other: biological examination at consultations at 3 and 6 months

INTERVENTIONS:
Other: biological examination at consultations at 3 and 6 months

SUMMARY:
The investigators set out to determine whether malnutrition delayed healing of foot lesions in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided oral consent
* Patients older than 18
* Patients with type 1 or 2 diabetes
* Patients who can be followed-up in the context of consultations for diabetic foot at the endocrinology, diabetology and metabolic diseases unit of Dijon CHU.
* Lesion situated on a toe or on the plantar or dorsal side of the foot
* Lesion that has evolved for 1 to 24 months

Exclusion Criteria:

* Adult under guardianship
* Patient without national health insurance
* Pregnant or breast-feeding women
* Patients with progressive cancer
* Patients with terminal renal insufficiency on dialysis
* Patient with severe respiratory insufficiency
* Patients with terminal heart failure
* Patients with severe liver failure
* Patients with immunodepriession (treatement with immunosuppressants, long-term corticotherapy, diseases leading to immunodepression)
* Patients with nephrotic syndrome (hypoalbuminemia)
* Patientswith a chronic inflammatory syndrome
* Alcohol consumption greater than 4 glasses per day
* Systemic infection uncontrolled by antibiotics
* Infected lesion with systemic repercussions
* Charcot foot
* Patients taking part or who have planned to take part in another clinical trial
* Severe disease affecting survival in the short term
* Lesion on an amputation
* Lesion of the ankle or leg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or 2 diabetes who have a lesion situated on a toe or on the plantar or dorsal side of the foot
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Percentage of healed lesions | After 24 weeks of follow-up

SECONDARY OUTCOMES:
Number of malnourished patients according to HAS 2003 and 2007 criteria | At inclusion

OTHER OUTCOMES:
Percentage of healed lesions during the follow-up | At 2, 4, 8, 12, 16 and 20 weeks
Number of malnourished patients at 12 and 24 weeks | At 12 and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Rouland A, Fourmont C, Sberna AL, Aho Glele LS, Mouillot T, Simoneau I, Verges B, Petit JM, Bouillet B. Malnutrition in type 2 diabetic patients does not affect healing of foot ulcers. Acta Diabetol. 2019 Feb;56(2):171-176. doi: 10.1007/s00592-018-1233-9. Epub 2018 Oct 3. PMID 30284047